CLINICAL TRIAL: NCT06629298
Title: Immediate Effects of Stochastic Whole-body Vibration Training on Balance and Executive Functions: A Randomized Controlled Trial
Brief Title: Effects of Stochastic Whole-body Vibration Training on Balance and Executive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2019-07-00005
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: One Experimental Group and one Control Group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 Hertz Whole-Body Vibration Intervention (Experimental): Three 1-minute sessions of stochastic whole-body vibration (SR-WBV) training with 1-minute breaks at 5 Hz
  Interventions: Other: 5Hz Stochastic Resonance Whole-Body Vibration Training
- 2 Hertz Whole-Body Vibration Intervention (Sham Comparator): Three 1-minute sessions of stochastic whole-body vibration (SR-WBV) training with 1-minute breaks at 2 Hz
  Interventions: Other: 2 Hz Stochastic Resonance Whole-Body Vibration Training

INTERVENTIONS:
Other: 5Hz Stochastic Resonance Whole-Body Vibration Training — Both the experimental group and the control group performed their training on an SRT Zeptor® Medical plus noise device (Frei Swiss AG, Zurich). The device featured two independent foot plates that vibrated stochastically in all three dimensions, resulting in multidimensional movement. During the training, participants were instructed to stand on the foot plates with both feet, keep their arms relaxed at their sides, maintain a slight bend in their knees, and focus their gaze on a fixation cross on the wall. Following the protocol used in Faes et al. (2018), each training session consisted of three series, each comprising one minute of vibration training followed by one minute of rest.
  The vibration frequency for the intervention group was set at 5 Hz.
  Arms: 5 Hertz Whole-Body Vibration Intervention
Other: 2 Hz Stochastic Resonance Whole-Body Vibration Training — Both the experimental group and the control group performed their training on an SRT Zeptor® Medical plus noise device (Frei Swiss AG, Zurich). The device featured two independent foot plates that vibrated stochastically in all three dimensions, resulting in multidimensional movement. During the training, participants were instructed to stand on the foot plates with both feet, keep their arms relaxed at their sides, maintain a slight bend in their knees, and focus their gaze on a fixation cross on the wall. Following the protocol used in Faes et al. (2018), each training session consisted of three series, each comprising one minute of vibration training followed by one minute of rest.
  The vibration frequency for the intervention group was set at 2 Hz.
  Arms: 2 Hertz Whole-Body Vibration Intervention

SUMMARY:
Falls represent a significant financial burden, costing millions of dollars annually in Switzerland (SUVA, 2022). Good cognitive abilities and good balance represent modifiable protective factors against falls (Kurz, 2008). The present study investigates the impact of stochastic whole-body vibration training (SR-WBV) on executive functions and balance. To this end, participants were randomized into an intervention group or a control group. Participants in the intervention group underwent SR-WBV at a frequency of 5 Hertz (Hz), while participants in the control group underwent SR-WBV at 2 Hz. The training on an SRT Zeptor® Medical plus noise device consisted of three one-minute intervals of vibration, interspersed with one-minute rest periods. Data on executive functions (Updating, Shifting, Inhibition) and balance were collected before and after the intervention , complemented by subjective assessments of concentration and balance through questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Pregnancy
* The presence of osteosynthetic materials (e.g., screws, plates, wires)
* Joint problems (particularly in the knees, hips, and back)
* Musculoskeletal issues
* Disc herniation
* Rheumatism
* Cardiovascular problems
* Balance disorders
* Red-green color blindness
* Intensive training within 24 hours prior to the assessment.
* Use of central nervous system medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Sense of Balance (Change from Baseline) | 19 min before and 19 min after the intervention (immediate effects)
  Measured with subjective scale (sense of balance from 0 to 10)
  How do you assess your personal sensations regarding muscles and joints (back pain, shoulder and neck pain, leg muscle pain, etc.) at this moment?
  Please slide the scale for each aspect to the most appropriate level.
  0 means no pain, and 10 means the most intense pain imaginable.
Balance (Change from Baseline) | Immediately before and 13 min after the intervention (immediate effects)
  Measured with the modified star excursion balance test (m-SEBT). Higher values indicate better balance with 0cm being the minimum and ca. 100cm indicating very good balance, i.e. reach distance.
  In this balance test, participants stand on one leg, while the range of motion of the other leg is measured in eight directions: anterior (ANT), posteromedial (PM), and posterolateral (PL).
  (Duration: 5 min)

SECONDARY OUTCOMES:
Executive functions (Shifting) (Change from Baseline) | 10 min before and 8 min after the intervention (immediate effects)
  Measured with the Trail-Making Test B
  For TMT B, participants were presented with circles filled with both numbers and letters. They were required to click the circles in ascending order, alternating between numbers and letters (e.g., 1, A, 2, B, 3, C). The practice task consisted of six circles, and the main test involved 24 circles. The processing time was measured in milliseconds.
  Thus, higher scores in the Trail-Making Test B indicate lower shifting ability.
  (Duration: 3 min)
Executive functions (Updating) (Change from Baseline) | 18 min before and immediately after the intervention (immediate effects)
  Measured with the Running Span-Task
  Participants were presented with a series of letters of varying lengths (3 to 8 letters).
  For each participant, both the total Running Span (sum of all correctly recalled target items) and the Running Span Score (sum of correctly recalled target items from sets that included at least one distractor) were calculated.
  Thus, higher scores (MIN = 0) in the Running Span-Task indicate higher updating ability.
  (Duration: 8 min)
Executive functions (Inhibition) (Change from Baseline) | 7 min before and 11 min after the intervention (immediate effects)
  Measured with the Stroop Test in milliseconds (Reaction Time)
  The reaction times (in milliseconds) for all correctly identified incongruent items were subtracted from those for control items.
  0 ms indicate no cognitive interference, i.e. maximal inhibitory control
  Thus, higher scores in the Stroop Test indicate higher cognitive interference, i.e. poorer inhibitory control
  (Duration: 2 min)

CONTACTS AND LOCATIONS:
Overall Officials: Achim Elfering, Prof. Dr. phil. nat., Study Chair — University of Bern
Locations (1):
- Institut für Psychologie, Arbeits- und Organisationspsychologie, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
Upon arrival, participants generated an individual ID, which was linked to their identity in a password-protected file for two weeks, during which they could request data deletion. After this period, the link was permanently removed, ensuring full anonymity. Only aggregated statistical analyses were conducted.

REFERENCES:
- [Background] Faes Y, Rolli Salathe C, Herlig ML, Elfering A. Beyond physiology: Acute effects of side-alternating whole-body vibration on well-being, flexibility, balance, and cognition using a light and portable platform A randomized controlled trial. Front Sports Act Living. 2023 Jan 30;5:1090119. doi: 10.3389/fspor.2023.1090119. eCollection 2023. PMID 36793620